CLINICAL TRIAL: NCT04158908
Title: Giving Information Systematically and Transparently in Lung and GI Cancer
Brief Title: Giving Information Systematically and Transparently in Lung and GI Cancer Phase 1
Acronym: Oncolo-GIST
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-07020392-Phase1; R21NR018693-01 (NIH)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Critical Illness; Oncology; Communication
MeSH Terms: conditions — Critical Illness; Neoplasms; Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oncolo-GIST Arm: Caregivers: Caregiver stakeholders were bereaved family members of a patient who had died from solid tumor cancer in the past year. Stakeholders reviewed an initial version of the Oncolo-GIST manual to provide feedback and refine the manual for Phase 2.
  Interventions: Behavioral: Oncolo-GIST
- Oncolo-GIST Arm: Clinicians: Clinician stakeholders were physicians, nurses, nurse practitioners, and social workers with expertise in treating advanced cancer patients. Stakeholders reviewed an initial version of the Oncolo-GIST manual to provide feedback and refine the manual for Phase 2.
  Interventions: Behavioral: Oncolo-GIST

INTERVENTIONS:
Behavioral: Oncolo-GIST — Oncolo-GIST is a brief, manualized communication intervention that guides oncologists in "gist communication" by itemizing 4 key steps in the process of imparting prognostic information.
  Topic covered include:
  1. Principles of introducing prognosis in the setting of worsened scan results
  2. Coupling communicating realistic prognoses with psychological support (e.g., saying "average life-expectancy is months…" with emphasizing that the oncology team "will always provide care for you")
  3. Addressing informational needs and psychological reactions
  4. Applying proven techniques for supporting patients who are reluctant to discuss prognosis.
  The 4-step guide will include brief video-clips of demonstrating each "talking point" with a standardized patient, including ideal scenarios, common pitfalls to avoid, and how to respond to patient reactions that are particularly challenging, such as responding to optimism, death anxiety, and reliance on faith.

SUMMARY:
When advanced disease progresses, there comes a time when an oncologists must explain to their patients that they only have months left to live. During these discussions the oncologist attempts to explain to the patient their prognoses and what it means for them going forward. However the investigator's prior studies shown that even when patients only have months left to live, most do not understand that their cancer is incurable and that it is late/end-stage.

Dying cancer patients who fully understand their prognosis are able to make more informed decisions and are therefore more likely to engage in advanced care planning, and receive care what in consistent with their values and preferences. They are also in a better position to avoid burdensome, non-beneficial care. The investigator developed Oncolo-GIST in order to help increase the number of patients who fully understand their prognosis and its implications.

Oncolo-GIST is an intervention aimed at enhancing clinicians' communication with patients by teaching them to relay information both sensitively and using simple terminology. The Oncolo-GIST training will provide instruction in areas such as how to introduce the topic of prognosis (describe scan results as "worse"), how to phrase the prognosis itself ("likely months, not years"), how to explain expected treatment outcomes (e.g., "not expected to be cured by treatment") and how to describe expected treatments impact on quality of life - that is, whether the anticancer treatment is likely to make them feel overall better or worse. The training materials consist of a manual and a set of videos that act out situations described in the manual.

The first phase of this study will consists of two parts:

1. Stakeholder Interviews: The investigator will obtain feedback from relevant stakeholders/key informants on Oncolo-GIST Version 1.0 manual and videos using a version of the Delphi method in which the investigator will interview bereaved family caregivers of advanced cancer patients (n=10) and oncology clinicians who care for patients with advanced gastrointestinal (GI) and thoracic (lung) cancers (n=10). The information gathered will be used to develop Oncolo-GIST Version 2.0.
2. Open Trial: The investigator will conduct an initial open trial of the Oncolo-GIST intervention to 10 advanced cancer patients (N=10) by participant clinicians (n=8). This will help us gather information about the feasibility and acceptability of the intervention to patients and oncologists and also inform changes for Oncolo-GIST Version 2.0.

This phase will be followed by second phased (listed in a separate record in ClinicalTrials.gov) that will include a randomized controlled trial of Oncolo-GIST Version 2.0. The record is titled "Giving Information Systematically and Transparently in Lung and GI Cancer Phase 2" and its NCT ID# isNCT04179305.

DETAILED DESCRIPTION:
Despite exciting recent advances in cancer treatments, there still, ultimately, comes a time when advanced disease progresses, and patients can reliably be expected to have months, not years, left to live. For patients with metastatic cancers studied in the investigator's Coping with Cancer NCI R01s, this comes after progression on 1st- or 2nd-line therapy -- be it chemo-, immune-, or targeted therapy. Prior studies conducted by the investigator have found that oncologists can reliably predict when patients have only months to live (e.g., remarkable agreement between oncologist estimates of months to live shared with patients and patients' actual survival of months). By contrast, patients appear largely unaware of their prognosis. For example, 5% of patients a median of 5 months from death, accurately understood they had incurable, late/end-stage, terminal cancer, and likely only months to live. Dying cancer patients appear to lack the prognostic understanding needed to make informed choices.

Patients who grasp that they are dying (e.g., the 8.6% who "get the gist" that they likely have months to live), relative to those who do not, have been shown to have: a) higher rates of advance care planning (ACP), b) receive less burdensome, unbeneficial care (e.g., fewer intensive care unit, ICU, stays, less cardiopulmonary resuscitation, CPR), and c) more value-consistent care. The investigator has found that patient prognostic understanding is improved by oncologist discussions of life-expectancy, but despite 71% of patients wanting to discuss prognosis with their oncologists (83% adult cancer patients thought prognostic information was extremely/very important), only 17.6% of cancer patients within months of death reported that they had discussed prognosis with their oncologist. Not only do oncologists appear to discuss prognosis less than patients want them to, but even when prognostic discussions do occur, the investigator has found that some approaches (e.g., matter-of-fact) are more effective than others (e.g., vague) for promoting patients' prognostic understanding. Thus, prior work identifies a need to improve communication to promote patient prognostic understanding in a way that oncologists will likely learn, accept, use, and possibly implement more broadly in clinical practice.

To address this need, the investigator developed the "Giving Information Simply &Transparently" (GIST), Oncolo-GIST intervention -- a manualized oncologist communication intervention that simplifies how to impart prognostic information by focusing on 4 basic steps: 1) Giving scan information, 2) Informing prognosis, 3) Strategizing sensitively, and 4) Transparently asking what the patient heard. Unlike traditional emphasis on numerical or medical details, the Oncolo-GIST approach is based on Reyna's Fuzzy-Trace Theory of decision-making, which emphasizes the need for an understanding of the bottom-line gist of a situation. The Oncolo-GIST approach distills prognostic discussions to clear communication of end-of-life (EoL) decision-making essentials (e.g., life-expectancy). 3 specific aims of the Oncolo-GIST approach will be tested in 2 phases:

Phase 1 will consist of two parts: 1) An interview of key stakeholders/key informants regarding Oncolo-GIST Version 1.0 in order to inform refinements to produce Oncolo-GIST Version 2.0. 2) An open trial of Oncolo-GIST Version 1.0 to inform refinements to produce Oncolo-GIST Version 2.0.

Phase 2 will involve a cluster randomized trial of Oncolo-GIST Version 2.0 on 50 patients with metastatic cancers worse on at least 1 line of therapy (chemo-, immune-, targeted), whose oncologists do not expect to survive 12 months. Patients will be assessed in the week prior to their scheduled scan, within 1 week of the clinic visit in which progressive scan results are discussed, and then 2 and 4 months later to explore intervention effects on primary and secondary outcomes, respectively. Oncologists will be assessed in the week following that same clinic visit to obtain their impressions of the discussion of prognosis and the patient's prognostic understanding.

In the phase one stakeholder interviews the investigator aims to obtain feedback on Oncolo-GIST Version 1.0 from stakeholders/key informants on an early draft of the Oncolo-GIST manual and proposed approach using a version of the Delphi method in which the investigator will interview bereaved family caregivers of advanced cancer patients (n=10) and oncology clinicians who care for patients with advanced gastrointestinal (GI) and thoracic (lung) cancers (n=10).

The Delphi method involves gathering opinions from "experts" (i.e., key informants/stakeholders), keeping feedback anonymous, and circulating it back to experts until consensus is reached. Two feedback rounds will occur in Phase 1. The investigator will recruit 10 bereaved caregivers (e.g., family/friends such as widows) of patients who died in the past year with primary diagnoses of GI or lung cancers, and 10 oncology clinicians (oncologists, palliative care physicians, nurses, nurse practitioners, social workers and psychologists) who care for patients with metastatic GI and lung cancers to obtain their feedback on the Oncolo-GIST Version 1.0 manual and procedures. Consenting subjects will be provided a copy of the Oncolo-GIST 4-step manual and a survey to obtain structured feedback on content, format, and language, which they will be asked to return within 4-6 weeks. Responses will be reviewed and compiled and returned to experts for additional feedback on the revised manual. A 30-60-minute follow-up telephone or video-conferenced interview of experts will be conducted by study staff within the following 2 weeks to identify important themes that may be clinically useful to incorporate into the Oncolo-GIST 2.0 intervention. Interviews will be audio-recorded, transcribed, and kept confidential. The investigator has successfully employed these procedures in a prior study, the EMPOWER intervention, with cancer patient caregivers (CA218313).

In the phase 1 open trial the investigator aims to determine feasibility and acceptability of Oncolo-GIST Version 1.0 in a trial of 10 advanced cancer patients to gather information of the feasibility and acceptability of the intervention to patients and oncologists and to inform refinements that will result in Version 2.0.

We will consent the 8 available oncologists identified by Drs. Shah and Saxena in the GI and lung cancer clinics at Weill Cornell Medicine (WCM). The PI will assign a number to each of the 8 oncologists and provide these numbers to the study statistician who will then randomly assign 4 of the numbers to training in the Oncolo-GIST intervention and the other 4 to usual care. Ten patients who meet the eligibility criteria will receive care from 1 of the 4 oncologists trained in the intervention. Phase 1 expert data will be reviewed and summarized, indicating strengths and weaknesses of the intervention and recommended modifications. Phase 1 open trial data will be cleaned, collated, and analyzed. Feasibility of patient recruitment and retention and oncologists' ability to apply the technique will be evaluated. Acceptability will be assessed among oncologists randomized to the intervention and their patients. The quantitative and qualitative data will inform refinements to the study design and intervention procedures that will result in Oncolo-GIST Version 2.0. A summary document will identify the main thematic issues raised in gathering of the Phase 1 data and will explain how they will (or why they will not) be addressed in revisions to the intervention. The 4 oncologists trained in Version 1.0 will receive additional instruction to be compliant with Version 2.0.

The details for Phase 2 are enumerated in a separate record marked "Giving Information Systematically and Transparently in Lung and GI Cancer Phase 2" (Oncolo-GIST P2), under NCT ID# NCT04179305.

ELIGIBILITY:
Clinicians (Stakeholder Interviews)

Inclusion Criteria:

* Currently care for patients with metastatic GI and lung cancers as an oncologist, palliative care physician, nurse, nurse practitioner, social worker, or psychologist

Exclusion Criteria:

* Does not currently care for patients with metastatic GI and lung cancers as either an oncologist, palliative care physician, nurse, nurse practitioner, social worker, or psychologist

Caregivers (Stakeholder Interviews)

Inclusion Criteria:

* Caregivers of patients who died in the past year with a primary diagnoses of GI or lung cancer

Exclusion Criteria:

* Caregivers of patients who died longer than 1 year from the time of enrollment
* Caregivers of a patient that did not have a primary diagnoses of GI or lung cancer
* Not fluent in English

Clinicians (Open Trial)

Inclusion Criteria:

* Specialize in Lung and GI cancers
* Currently provide care at the WCM Lung and GI cancer clinics
* Fluent in English

Exclusion Criteria:

* Does not specialize in Lung and GI cancers
* Does not currently provide care at the WCM Lung and GI cancer clinics
* Not fluent in English

Patients (Open Trial)

Inclusion Criteria:

* Receiving ongoing care (≥ 2 visits) that includes regular scans
* Progression on at least 1 line of systemic cancer therapy
* Prognosis from an oncologist of less than 12 months
* Receiving care from an oncologist participating in the Oncolo-GIST study
* Fluent in English

Exclusion Criteria:

* Does not specialize in Lung and GI cancers
* Does not currently provide care at the WCM Lung and GI cancer clinics
* Not fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caregivers were selected from among families of past patients identified by clinicians at Weill Cornell Medicine. Clinicians with expertise in palliative medicine were selected from among colleagues of PI.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly G Prigerson, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambden J, Zhang B, Friedlander R, Prigerson HG. Accuracy of Oncologists' Life-Expectancy Estimates Recalled by Their Advanced Cancer Patients: Correlates and Outcomes. J Palliat Med. 2016 Dec;19(12):1296-1303. doi: 10.1089/jpm.2016.0121. Epub 2016 Aug 30. PMID 27574869
- [Background] Enzinger AC, Zhang B, Schrag D, Prigerson HG. Outcomes of Prognostic Disclosure: Associations With Prognostic Understanding, Distress, and Relationship With Physician Among Patients With Advanced Cancer. J Clin Oncol. 2015 Nov 10;33(32):3809-16. doi: 10.1200/JCO.2015.61.9239. Epub 2015 Oct 5. PMID 26438121
- [Background] Epstein AS, Prigerson HG, O'Reilly EM, Maciejewski PK. Discussions of Life Expectancy and Changes in Illness Understanding in Patients With Advanced Cancer. J Clin Oncol. 2016 Jul 10;34(20):2398-403. doi: 10.1200/JCO.2015.63.6696. Epub 2016 May 23. PMID 27217454
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Wright AA, Zhang B, Keating NL, Weeks JC, Prigerson HG. Associations between palliative chemotherapy and adult cancer patients' end of life care and place of death: prospective cohort study. BMJ. 2014 Mar 4;348:g1219. doi: 10.1136/bmj.g1219. PMID 24594868
- [Background] Prigerson HG. Socialization to dying: social determinants of death acknowledgement and treatment among terminally ill geriatric patients. J Health Soc Behav. 1992 Dec;33(4):378-95. PMID 1464721
- [Background] Wright AA, Zhang B, Ray A, Mack JW, Trice E, Balboni T, Mitchell SL, Jackson VA, Block SD, Maciejewski PK, Prigerson HG. Associations between end-of-life discussions, patient mental health, medical care near death, and caregiver bereavement adjustment. JAMA. 2008 Oct 8;300(14):1665-73. doi: 10.1001/jama.300.14.1665. PMID 18840840
- [Background] Mack JW, Fasciano KM, Block SD. Communication About Prognosis With Adolescent and Young Adult Patients With Cancer: Information Needs, Prognostic Awareness, and Outcomes of Disclosure. J Clin Oncol. 2018 Jun 20;36(18):1861-1867. doi: 10.1200/JCO.2018.78.2128. Epub 2018 Apr 23. PMID 29683788
- [Background] Reyna VF. Theories of medical decision making and health: an evidence-based approach. Med Decis Making. 2008 Nov-Dec;28(6):829-33. doi: 10.1177/0272989X08327069. No abstract available. PMID 19020341
- [Background] Elsayyad A. Informed consent for comparative effectiveness trials. N Engl J Med. 2014 May 15;370(20):1958-9. doi: 10.1056/NEJMc1403310. No abstract available. PMID 24827054
- [Background] Spellecy R, Tarima S, Denzen E, Moore H, Abhyankar S, Dawson P, Foley A, Gersten I, Horwitz M, Idossa L, Joffe S, Kamani N, King R, Lazaryan A, Morris L, Horowitz MM, Majhail NS. Easy-to-Read Informed Consent Form for Hematopoietic Cell Transplantation Clinical Trials: Results from the Blood and Marrow Transplant Clinical Trials Network 1205 Study. Biol Blood Marrow Transplant. 2018 Oct;24(10):2145-2151. doi: 10.1016/j.bbmt.2018.04.014. Epub 2018 Apr 18. PMID 29679770
- [Background] Tulsky JA, Arnold RM, Alexander SC, Olsen MK, Jeffreys AS, Rodriguez KL, Skinner CS, Farrell D, Abernethy AP, Pollak KI. Enhancing communication between oncologists and patients with a computer-based training program: a randomized trial. Ann Intern Med. 2011 Nov 1;155(9):593-601. doi: 10.7326/0003-4819-155-9-201111010-00007. PMID 22041948
- [Background] Mitchell SL, Shaffer ML, Cohen S, Hanson LC, Habtemariam D, Volandes AE. An Advance Care Planning Video Decision Support Tool for Nursing Home Residents With Advanced Dementia: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2018 Jul 1;178(7):961-969. doi: 10.1001/jamainternmed.2018.1506. PMID 29868778
- [Background] Epstein AS, Volandes AE, Chen LY, Gary KA, Li Y, Agre P, Levin TT, Reidy DL, Meng RD, Segal NH, Yu KH, Abou-Alfa GK, Janjigian YY, Kelsen DP, O'Reilly EM. A randomized controlled trial of a cardiopulmonary resuscitation video in advance care planning for progressive pancreas and hepatobiliary cancer patients. J Palliat Med. 2013 Jun;16(6):623-31. doi: 10.1089/jpm.2012.0524. Epub 2013 Apr 22. PMID 23725233
- [Background] Reyna VF. A theory of medical decision making and health: fuzzy trace theory. Med Decis Making. 2008 Nov-Dec;28(6):850-65. doi: 10.1177/0272989X08327066. Epub 2008 Nov 17. PMID 19015287
- [Background] Derry HM, Maciejewski PK, Epstein AS, Shah MA, LeBlanc TW, Reyna V, Prigerson HG. Associations between Anxiety, Poor Prognosis, and Accurate Understanding of Scan Results among Advanced Cancer Patients. J Palliat Med. 2019 Aug;22(8):961-965. doi: 10.1089/jpm.2018.0624. Epub 2019 Feb 6. PMID 30724692
- [Background] Fenton JJ, Duberstein PR, Kravitz RL, Xing G, Tancredi DJ, Fiscella K, Mohile S, Epstein RM. Impact of Prognostic Discussions on the Patient-Physician Relationship: Prospective Cohort Study. J Clin Oncol. 2018 Jan 20;36(3):225-230. doi: 10.1200/JCO.2017.75.6288. Epub 2017 Nov 17. PMID 29148892
- [Background] de Meyrick J: The Delphi Method and Health Research. Health Education 103:7-16, 2003
- [Background] Bell ML, Whitehead AL, Julious SA. Guidance for using pilot studies to inform the design of intervention trials with continuous outcomes. Clin Epidemiol. 2018 Jan 18;10:153-157. doi: 10.2147/CLEP.S146397. eCollection 2018. PMID 29403314
- [Background] Reyna VF, Nelson WL, Han PK, Pignone MP. Decision making and cancer. Am Psychol. 2015 Feb-Mar;70(2):105-18. doi: 10.1037/a0036834. PMID 25730718
- [Background] Singh S, Cortez D, Maynard D, Cleary JF, DuBenske L, Campbell TC. Characterizing the Nature of Scan Results Discussions: Insights Into Why Patients Misunderstand Their Prognosis. J Oncol Pract. 2017 Mar;13(3):e231-e239. doi: 10.1200/JOP.2016.014621. Epub 2017 Jan 17. PMID 28095172
- [Background] Shen MJ, Trevino KM, Prigerson HG. The interactive effect of advanced cancer patient and caregiver prognostic understanding on patients' completion of Do Not Resuscitate orders. Psychooncology. 2018 Jul;27(7):1765-1771. doi: 10.1002/pon.4723. Epub 2018 Apr 30. PMID 29611241
- [Background] Kurita K, Siegler EL, Reid MC, Maciejewski RC, Prigerson HG. It Is Not What You Think: Associations Between Perceived Cognitive and Physical Status and Prognostic Understanding in Patients With Advanced Cancer. J Pain Symptom Manage. 2018 Aug;56(2):259-263. doi: 10.1016/j.jpainsymman.2018.04.016. Epub 2018 May 10. PMID 29753102
- [Background] Cohen SM, Maciejewski RC, Shah MA, Trevino KM, Shen MJ, Maciejewski PK, Prigerson HG. Being present: oncologists' role in promoting advanced cancer patients' illness understanding. Cancer Med. 2018 Apr;7(4):1511-1518. doi: 10.1002/cam4.1389. Epub 2018 Feb 26. PMID 29479843
- [Background] Morse JM: Designing funded qualitative research. Handbook of qualitative research, Denzin and Lincoln (eds), Thousand Oaks, CA, Sage Publications, Inc:220-235, 1994
- [Background] Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975 Oct;23(10):433-41. doi: 10.1111/j.1532-5415.1975.tb00927.x. PMID 1159263
- [Background] van Vliet LM, Epstein AS. Current state of the art and science of patient-clinician communication in progressive disease: patients' need to know and need to feel known. J Clin Oncol. 2014 Nov 1;32(31):3474-8. doi: 10.1200/JCO.2014.56.0425. Epub 2014 Sep 29. No abstract available. PMID 25267758
- [Background] Gilligan T, Coyle N, Frankel RM, Berry DL, Bohlke K, Epstein RM, Finlay E, Jackson VA, Lathan CS, Loprinzi CL, Nguyen LH, Seigel C, Baile WF. Patient-Clinician Communication: American Society of Clinical Oncology Consensus Guideline. J Clin Oncol. 2017 Nov 1;35(31):3618-3632. doi: 10.1200/JCO.2017.75.2311. Epub 2017 Sep 11. PMID 28892432
- [Background] Back AL, Arnold RM. Discussing prognosis: "how much do you want to know?" talking to patients who are prepared for explicit information. J Clin Oncol. 2006 Sep 1;24(25):4209-13. doi: 10.1200/JCO.2006.06.007. No abstract available. PMID 16943539
- [Background] Hagerty RG, Butow PN, Ellis PM, Lobb EA, Pendlebury SC, Leighl N, MacLeod C, Tattersall MH. Communicating with realism and hope: incurable cancer patients' views on the disclosure of prognosis. J Clin Oncol. 2005 Feb 20;23(6):1278-88. doi: 10.1200/JCO.2005.11.138. PMID 15718326
- [Background] Jacobsen J, Brenner K, Greer JA, Jacobo M, Rosenberg L, Nipp RD, Jackson VA. When a Patient Is Reluctant To Talk About It: A Dual Framework To Focus on Living Well and Tolerate the Possibility of Dying. J Palliat Med. 2018 Mar;21(3):322-327. doi: 10.1089/jpm.2017.0109. Epub 2017 Oct 3. PMID 28972862
- [Background] McCambridge J, Witton J, Elbourne DR. Systematic review of the Hawthorne effect: new concepts are needed to study research participation effects. J Clin Epidemiol. 2014 Mar;67(3):267-77. doi: 10.1016/j.jclinepi.2013.08.015. Epub 2013 Nov 22. PMID 24275499
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of health care interventions: A theoretical framework and proposed research agenda. Br J Health Psychol. 2018 Sep;23(3):519-531. doi: 10.1111/bjhp.12295. Epub 2018 Feb 16. No abstract available. PMID 29453791
- [Background] Cohen SR, Mount BM, Strobel MG, Bui F. The McGill Quality of Life Questionnaire: a measure of quality of life appropriate for people with advanced disease. A preliminary study of validity and acceptability. Palliat Med. 1995 Jul;9(3):207-19. doi: 10.1177/026921639500900306. PMID 7582177
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Wright AA, Mack JW, Kritek PA, Balboni TA, Massaro AF, Matulonis UA, Block SD, Prigerson HG. Influence of patients' preferences and treatment site on cancer patients' end-of-life care. Cancer. 2010 Oct 1;116(19):4656-63. doi: 10.1002/cncr.25217. PMID 20572030
- [Background] Phillips RS, Wenger NS, Teno J, Oye RK, Youngner S, Califf R, Layde P, Desbiens N, Connors AF Jr, Lynn J. Choices of seriously ill patients about cardiopulmonary resuscitation: correlates and outcomes. SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Am J Med. 1996 Feb;100(2):128-37. doi: 10.1016/s0002-9343(97)89450-8. PMID 8629646
- [Background] Mack JW, Block SD, Nilsson M, Wright A, Trice E, Friedlander R, Paulk E, Prigerson HG. Measuring therapeutic alliance between oncologists and patients with advanced cancer: the Human Connection Scale. Cancer. 2009 Jul 15;115(14):3302-11. doi: 10.1002/cncr.24360. PMID 19484795
- [Background] Davis TC, Long SW, Jackson RH, Mayeaux EJ, George RB, Murphy PW, Crouch MA. Rapid estimate of adult literacy in medicine: a shortened screening instrument. Fam Med. 1993 Jun;25(6):391-5. PMID 8349060
- [Background] Balboni TA, Prigerson HG, Balboni MJ, Enzinger AC, VanderWeele TJ, Maciejewski PK. A scale to assess religious beliefs in end-of-life medical care. Cancer. 2019 May 1;125(9):1527-1535. doi: 10.1002/cncr.31946. Epub 2019 Mar 2. PMID 30825390
- [Background] Canner PL. Covariate adjustment of treatment effects in clinical trials. Control Clin Trials. 1991 Jun;12(3):359-66. doi: 10.1016/0197-2456(91)90016-f. PMID 1651207
- [Background] Begg C, Cho M, Eastwood S, Horton R, Moher D, Olkin I, Pitkin R, Rennie D, Schulz KF, Simel D, Stroup DF. Improving the quality of reporting of randomized controlled trials. The CONSORT statement. JAMA. 1996 Aug 28;276(8):637-9. doi: 10.1001/jama.276.8.637. No abstract available. PMID 8773637
- [Background] Grant S, Mayo-Wilson E, Montgomery P, Macdonald G, Michie S, Hopewell S, Moher D; , on behalf of the CONSORT-SPI Group. CONSORT-SPI 2018 Explanation and Elaboration: guidance for reporting social and psychological intervention trials. Trials. 2018 Jul 31;19(1):406. doi: 10.1186/s13063-018-2735-z. PMID 30060763
- [Background] Schafer JL, Olsen MK. Multiple Imputation for Multivariate Missing-Data Problems: A Data Analyst's Perspective. Multivariate Behav Res. 1998 Oct 1;33(4):545-71. doi: 10.1207/s15327906mbr3304_5. PMID 26753828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians
Started | 11 | 9
Completed | 10 | 8
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 8 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Education [Count of Participants; unit: Participants]
  High School | 1 | 0 | 1
  Some College | 1 | 0 | 1
  College | 4 | 1 | 5
  Postgraduate | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Proposed Intervention According to a Structured Qualitative Survey of Caregivers
Description: Acceptability will be determined by requesting and comparing caregivers' responses to the specific phrasings indicated in the Oncolo-GIST manual for oncologists, with regard to sensitivity and comprehensibility.
Time Frame: From viewing the intervention to completing the survey, a period of approximately 2 hours occurring 1 week after enrollment.
Population: All caregivers who viewed and commented on the manual.
Measure: Count of Participants; unit: Participants
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians
Number analyzed (Participants) | 10 | 0
Participants
  Stakeholders found the intervention generally sensitive and empathetic. | 9 |
  Phrases such as "months, not years" are clear and though difficult, important for patients to hear. | 10 |
  "Prepare for the worst" may be overly harsh; noted and alternatives provided in new manual. | 1 |
  Some participants found oncologist's delivery in videos "cold" and advised showing more empathy. | 3 |

2. Primary Outcome: Acceptability of the Proposed Intervention According to a Structured Qualitative Survey of Clinicians
Description: Acceptability will be determined by requesting and comparing a range of clinicians' responses to the specific phrasings indicated in the Oncolo-GIST manual, with regard to sensitivity, comprehensibility, and accordance with the principles of informed consent.
Time Frame: as for outcome 1
Population: All clinicians who viewed and commented on the manual
Measure: Count of Participants; unit: Participants
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians
Number analyzed (Participants) | 0 | 8
Participants
  Generally very favorable reactions; respondents found intervention sensitive and empathetic. |  | 8
  Possible cultural insensitivity in asking how some patients feel after news; noted in manual. |  | 1
  Intervention may blur lines between physician and therapist; involve mental health professionals. |  | 2
  Some participants advised against breathing exercises in favor of therapeutic conversation. |  | 3

3. Primary Outcome: Feasibility of the Proposed Intervention According to a Structured Qualitative Survey of Clinicians
Description: Feasibility will be determined by requesting and comparing clinicians' responses to the manual's format and content, to determine the extent to which it is implementable in a clinical setting.
Time Frame: as for outcome 1
Population: All clinicians who viewed and remarked on the manual.
Measure: Count of Participants; unit: Participants
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians
Number analyzed (Participants) | 0 | 8
Participants
  Clinicians broadly found the intervention helpful, feasible, and implementable in clinical setting. |  | 8
  Some clinicians noted physicians (especially if older) could be resistant to training in a new style |  | 1
  Clinicians noted that time constraints would make some therapeutic aspects of intervention difficult |  | 2

4. Primary Outcome: Potential Improvements to the Oncolo-GIST Manual According to Structured Qualitative Surveys
Description: Using a version of the Delphi method 14, the responses of caregivers and clinicians will be anonymously amalgamated and compared in order to identify common criticisms of or suggestions for the manual, by frequency or priority, which can be implemented in Oncolo-GIST 2.0.
Time Frame: as for outcome 1
Population: All stakeholders who viewed and commented on the manual.
Measure: Count of Participants; unit: Participants
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians
Number analyzed (Participants) | 10 | 8
Participants
  Some participants advised improving manual videos to emphasize compassion and personability. | 3 | 1
  Teach-back elements in manual should be revised to be sensitive and avoid "quizzing" patients. | 1 | 1
  When training physicians, acceptability could be improved by framing O-Gist as a "time estimate" | 0 | 1
  The physician could give a brief overview of the disease course to orient the patient. | 1 | 0

ADVERSE EVENTS:
Time Frame: From viewing the intervention to completing the survey, a period of approximately 2 hours occurring 1 week after enrollment.
Description: For the purpose of this study, an AE is defined as a participant experiencing severe psychological distress, regardless of attribution. AEs are considered treatment-related if the participant's psychological distress can be probably or definitely be attributed to study activities (viewing the manual or completing study assessments). Serious adverse events (SAEs) were not monitored or assessed.
Arm/Group | Oncolo-GIST Arm: Caregivers | Oncolo-GIST Arm: Clinicians
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
Two participants (one clinician, one stakeholder) were unable to complete the study due to difficulties caused by COVID-19. In addition, racial and ethnic diversity among stakeholders was limited, which may have limited the study's ability to capture important cultural perspectives. Additionally, only three male caregivers participated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT04158908/Prot_SAP_000.pdf